CLINICAL TRIAL: NCT00755963
Title: The Influence of Hormone Replacement Therapy on the Cerebral Serotonin-1A Receptor Distribution and Mood in Postmenopausal Women
Brief Title: Effects of Hormone Replacement Therapy on the Serotonergic System and Mood in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: ao. Univ.-Prof. Dr. DDr.h.c. Siegfried Kasper, Department of Psychiatry and Psychotherapy, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PM-20070724; EudraCT: 2007-005685-12; EC 593/2007
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Hormone Replacement
MeSH Terms: interventions — Estradiol; Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: estradiol valerate; Drug: micronized progesterone
- 2 (Experimental)
  Interventions: Drug: estradiol valerate
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: estradiol valerate — Progynova® 21; 2mg/d
  Arms: 1; 2
Drug: micronized progesterone — Utrogestan®; 200mg/d
  Arms: 1
Drug: placebo — maltodextrin
  Arms: 3

SUMMARY:
Menopausal and postmenopausal women compose almost 20% of the Austrian population. Two thirds of all austrian women suffering from depression or anxiety disorders are over 45 years old. The serotonergic system, partially regulated by the steroid hormones estrogen and progesterone, plays a major role in the pathogenesis and treatment of these illnesses. To examine the effect of the hormone replacement therapy on the serotonergic system, twenty-four postmenopausal women will be measured using positron emission tomography (PET). The volunteers will participate in two PET scans. The first PET scan will be performed right before the hormone treatment starts, the second PET scan about 8 weeks after daily treatment with (1) a combination of estrogen and progesterone or (2) estrogen and placebo. This imaging study hypothesizes that the expression of the main inhibiting serotonergic receptor (the serotonin-1A receptor) will be altered by the hormone therapy. The results of the study might lead to new strategies in the treatment of psychiatric illnesses during and after the menopausal transition.

ELIGIBILITY:
Inclusion Criteria

* Postmenopausal females (over 14 months of amenorrhoea)
* Age 50 - 65 years
* Signed informed consent form
* Consent not to participate in PET or SPECT studies with an added equivalence dose of over 15 mSv within 10 years following the final assessment of the participant in this study

Exclusion criteria

* Steroid hormone treatment within 6 months prior to the inclusion
* Current substance abuse
* History of any malign illness
* Any implant or stainless steel graft
* Concomitant neurological illness
* Concomitant psychiatric disorder except anxiety disorders or depression
* Treatment with a psychotropic agent targeting serotonin-1A and serotonin-2A receptors or the serotonin transporter such as buspirone, pindolol or SSRIs
* Clinically relevant abnormalities in the general physical examination and the routine laboratory screening
* Concomitant major illness, especially: liver disease, disorders of the endocrine system, osteoporosis (when treated with vitamine D), any clinically relevant vascular or heart diseases
* One of the following gynaecological diseases: ovariectomy, hysterectomy, endometriosis, cervical smear test: PAP > II
* Failures to comply with the study protocol or to follow the instructions of the investigating team
* Investigations using PET or SPECT within 10 years prior to the inclusion

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Serotonin-1A receptor binding potential | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Siegfried Kasper, MD, Principal Investigator — Medical University of Vienna, Dept. of Psychiatry and Psychotherapy
Locations (1):
- Medical University of Vienna, Dept. of Psychiatry and Psychotherapy, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Kranz GS, Rami-Mark C, Kaufmann U, Baldinger P, Hahn A, Hoflich A, Savli M, Stein P, Wadsak W, Mitterhauser M, Winkler D, Lanzenberger R, Kasper S. Effects of hormone replacement therapy on cerebral serotonin-1A receptor binding in postmenopausal women examined with [carbonyl-(1)(1)C]WAY-100635. Psychoneuroendocrinology. 2014 Jul;45:1-10. doi: 10.1016/j.psyneuen.2014.03.004. Epub 2014 Mar 20. PMID 24845171